CLINICAL TRIAL: NCT01268553
Title: Transition From Parenteral Prostanoids to Inhaled Treprostinil
Brief Title: Transition From Injectable Prostacyclin Medication to Inhaled Prostacyclin Medication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, ronald oudiz, m.d., Professor of Medicine, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tyvaso Switch
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; inhaled prostacyclin
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active treatment (Experimental): This is the only arm in the trial. All enrolled subjects will be attempted to transition to inhaled treprostinil. There is no placebo and control arm.
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — Transition to inhaled treprostinil
  Other Names: Tyvaso

SUMMARY:
The purpose of this study is to assess tolerability and clinical effects of transition from intravenous (IV, needle in the vein) or subcutaneous (SQ, needle in the skin) to the recently-approved inhaled treprostinil (Tyvaso) for the treatment of pulmonary arterial hypertension (PAH).

Our hypothesis is that the transition to inhaled treprostinil will be tolerated by patients.

The intravenous and subcutaneous drugs epoprostenol and treprostinil received approval for treatment of PAH many years ago. While these medications improve exercise capacity and the symptoms of PAH, they are given by injection and thus have several side effects, such as pain and catheter infection. This has resulted in many patients either refusing to take the medication or quitting these medications because of not tolerating them.

The only other form of prostacyclin treatment available for PAH patients is inhaled. There are 2 inhaled prostacyclins approved for PAH, however one of these requires at least 6 inhalations per day, every day, and takes about 30 minutes to inhale each time. Thus, it has not been a regularly-used medication and issues surrounding compliance make it a riskier drug to use if patients do not get their full doses every day. The other inhaled medication, treprostinil, was approved a few months ago, only needs to be given 4 times a day, and takes about 2-3 minutes to inhale.

Since inhaled treprostinil can be administered easily, it is anticipated that many patients will transition from epoprostenol or treprostinil to the recently approved inhaled treprostinil, however we do not know if this is a safe or effective way to manage patients. Thus, the goal of this prospective study is to gather observational data regarding how that switch is made, tolerability of the switch, and, to the extent possible with this methodology, assess clinical effects of the switch.

This is a prospective study. Twenty patients > 18 years old with PAH will be enrolled. Patients enrolled will be those in whom a clinical decision to convert from either IV epoprostenol, IV treprostinil, or SQ treprostinil to inhaled treprostinil therapy has been made. This is usually the result of patients asking to switch to inhaled therapy, but only allowed by physicians if they feel the switch would be safe.

If eligible, and after informed consent, patients will have a history and physical examination, a 6 min walk test, a cardiopulmonary exercise test (CPET), blood tests, and a symptom questionnaire will be filled out. Patients will then be admitted to the hospital where a monitoring catheter will be placed inside the patient's heart and inhaled treprostinil will be initiated, while the dose of IV/SQ medication is reduced over about 24-26 hours.

Clinical follow-up will be at weeks 1, 4, and 12.

The procedures above are all part of the routine clinical care that patients would receive if they were to be transitioned to inhaled therapy, including the hospitalization and catheterization. The criteria for them to be able to be switched are conservative. Pressure in their heart and lungs must be low (mPAP < 40 mmHg and RAP <12 mmHg on catheterization), and their dose of IV or SQ medication must be low (< 20 ng/kg/min). Regarding the patient subset enrolled in this study in whom a clinical decision to convert transition therapy has been made, we will try to ensure that our clinical decision-making will not be influenced by the need to enroll subjects in the study by explicitly noting the potential for conflict of interest with each patient (addressed in the ICF). We will not make a clinical decision for our patients based on the desire to fill the study numbers, and every will be made to avoid the potential for a perceived conflict of interest.

DETAILED DESCRIPTION:
Purpose This study proposes to investigate the safety, tolerability, and feasibility of transitioning patients with PAH from intravenous or subcutaneous prostacyclin analogs to inhaled treprostinil using a defined protocol. Twenty-one patients from three PH specialty referral centers will be enrolled in this 12-week, prospective, open-label study. If subjects meet inclusion and exclusion criteria, they will be switched from intravenous or subcutaneous prostacyclin analogs to inhaled treprostinil according to a defined transition protocol.

Background Parenteral prostacyclin analogs improve exercise capacity and survival in patients with pulmonary arterial hypertension (PAH), however practical issues can limit their tolerability in some patients. The prostacyclin analogue treprostinil has been shown to improve exercise capacity and signs/symptoms of PAH, while delivered via four 2-3 minute inhalation periods per day. In addition, there is extensive worldwide experience with the subcutaneous and intravenous forms of treprostinil, with documented safety, efficacy, and tolerability.

Prior published studies have examined the feasibility of prostacyclin transitions, including transition from intravenous epoprostenol to non-parenteral PAH treatments, from subcutaneous to intravenous treprostinil, and from intravenous prostanoids to subcutaneous treprostinil.

There is currently no published experience examining the safety, tolerability and feasibility of transitioning patients from parenteral prostanoids to inhaled treprostinil.

ELIGIBILITY:
Inclusion Criteria:

* Patients with WHO group I PAH
* Stable patients with NYHA/WHO functional class I or II
* Age >18
* Treatment for PAH with parenteral prostanoid (IV epoprostenol, IV or SQ treprostinil) for at least 90 days
* Dose of prostanoid < 20 ng/kg/min
* mPAP < 40 mmHg and RAP <12 mmHg on catheterization
* Clinical decision to convert from parenteral prostanoid therapy to inhaled treprostinil therapy

Exclusion Criteria:

* Concomitant underlying medical condition limiting ability to perform exercise
* Addition of new PAH medication within the past 90 days prior to enrollment
* Participation in a clinical study involving an investigational drug or device < 4 weeks prior to the screening visit
* Any additional contraindications and precautions specified in the package inserts for treprostinil (Tyvaso) not listed above

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-08; Primary Completion 2016-10-05 (Actual); Study Completion 2016-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Oudiz, MD, Principal Investigator — LA Biomed
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - University of CA, San Francisco, San Francisco, California
  - Harbor-UCLA Medical Center, Torrance, California

REFERENCES:
- [Derived] Oudiz R, Agarwal M, Rischard F, De Marco T. An advanced protocol-driven transition from parenteral prostanoids to inhaled trepostinil in pulmonary arterial hypertension. Pulm Circ. 2016 Dec;6(4):532-538. doi: 10.1086/688711. PMID 28090295

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Single Arm Group: World Health Organization (WHO) group 1 PAH patients receiving long-term parenteral prostanoids
Period: Overall Study
Arm/Group | Open Label Single Arm Group
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Single Arm Group
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9
pulmonary vascular resistance [Mean (Standard Deviation); unit: Wood Units] — Population: 3 screen failures
  Wood Units
    number analyzed (Participants) | 6
    (all) | 4.2 (2.4)
6-minute walk distance [Mean (Standard Deviation); unit: meters] — Population: 3 screen failures
  meters
    number analyzed (Participants) | 6
    (all) | 334 (132)
peak oxygen consumption [Mean (Standard Deviation); unit: L/min] — Population: 3 screen failures
  L/min
    number analyzed (Participants) | 6
    (all) | 1.0 (0.2)
ratio of minute ventilation to CO2 output [Mean (Standard Deviation); unit: ratio] — Population: 3 screen failures
  ratio
    number analyzed (Participants) | 6
    (all) | 32 (2)
The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) [Mean (Standard Deviation); unit: units on a scale] — CAMPHOR is a questionnaire that measures quality of life of patients with pulmonary hypertension using units on a scale, 0-25, higher = worse Population: 3 screen failures
  units on a scale
    number analyzed (Participants) | 6
    (all) | 6.8 (6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Adverse Events
Description: The number of adverse events will be recorded at transition, 4 weeks, and 12 weeks.
Time Frame: 12 Weeks
Population: Number of patients weaned off of their parenteral prostanoids without adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Single Arm Group
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Number of Participants Without Clinical Worsening
Description: Clinical worsening is defined as any of the following:
  * All-cause mortality
  * Nonelective hospital stay for PAH (with predefined criteria, usually for initiation of intravenous prostanoids, lung transplantation, or septostomy)
  * Disease progression defined as a reduction from baseline in the 6MW test by 15%, confirmed by 2 studies done within 2 weeks plus worsening functional class
Time Frame: 12 weeks
Population: Patients weaned off of their parenteral prostanoids without Clinical Worsening
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Single Arm Group
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Change in 6-minute Walk Distance
Description: Change in 6-minute walk distance from baseline to 12 weeks.
Time Frame: 12 weeks
Population: Mean change in 6-minute walk distance
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Open Label Single Arm Group
Number analyzed (Participants) | 6
meters | 20 (58)

4. Secondary Outcome: VE/VCO
Description: Ventilatory efficiency measured with cardiopulmonary exercise testing
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Open Label Single Arm Group
Number analyzed (Participants) | 6
ratio | 1.2 (2.0)

5. Secondary Outcome: CAMPHOR: Cambridge Pulmonary Hypertension Outcome Review; Construct = Quality of Life
Description: The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) is a disease specific patient-reported outcome measure which assesses quality of life of patients with pulmonary hypertension (PH). QoL scores (total) range from 0-25, with higher scores indicating worse quality of life
Time Frame: 12 q=weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Single Arm Group
Number analyzed (Participants) | 6
units on a scale | -0.5 (3.4)

6. Secondary Outcome: N-terminal Pro BNP Level
Description: N-terminal pro BNP level
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Open Label Single Arm Group
Number analyzed (Participants) | 6
pg/mL | 14 (52)

ADVERSE EVENTS:
Arm/Group | Open Label Single Arm Group
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No